CLINICAL TRIAL: NCT05126745
Title: Assessment of Catheter Flow Direction Using Color Flow Doppler in Labor Epidurals: an Observational Study
Brief Title: Assessment of Catheter Flow Direction Using Color Flow Doppler in Labor Epidurals
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21-07
Record Dates: First submitted 2021-10-25; First posted 2021-11-19 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Labor Pain
Keywords: epidural catheter; epidural analgesia; labor epidural; ultrasound; Doppler
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who had an epidural placed for labour: Patients who had an epidural placed for labour may take part. Study procedures will take place after delivery and prior to removal of the epidural catheter.
  Interventions: Device: color flow Doppler ultrasonography

INTERVENTIONS:
Device: color flow Doppler ultrasonography — Doppler ultrasonography

SUMMARY:
Epidural analgesia is commonly used for pain relief in labor and involves placement of a catheter in the epidural space. Failure of epidural analgesia may occur in 12-16% of epidural catheter placements. It is defined as inadequate analgesia after the local anesthetic loading dose, despite use of appropriate dose/concentration of local anesthetic. Failure to provide adequate epidural analgesia is commonly caused by malposition of the epidural catheter. Many factors may influence the position of the tip of the epidural catheter and the resulting spread of local anesthetic into the epidural space, and consequently the quality of analgesia. Previously, X-ray exposure was required to assess catheter position in the epidural space. Recent developments have allowed the anesthesiologist to assess the catheter position at the bedside after its placement, using color flow Doppler ultrasonography.

The investigators will perform an observational study to determine epidural catheter flow direction in the obstetrical population using color flow Doppler ultrasound. Women who have delivered under epidural analgesia, either vaginal or caesarean delivery, will be approached for the study before the epidural catheter is removed.

The investigators aim to determine epidural flow relative to the insertion site, describe the findings and to correlate them with other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Women who have delivered under epidural analgesia
* Women who have vaginal or caesarean delivery
* Women with the epidural catheter still in place

Exclusion Criteria:

-Women who experience fetal or maternal complications during delivery

Ages: 18 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: Women who have delivered under epidural analgesia, either with vaginal or caesarean delivery, will be approached for the study before the epidural catheter is removed.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Visualization of flow relative to the interspace insertion level as assessed by color flow Doppler ultrasound | 15 min
  Visualization of flow relative to the interspace insertion level as assessed by color flow Doppler ultrasound (at insertion level [yes/no], above insertion level [yes/no], below insertion level [yes/no], no visualization of flow in any space).

SECONDARY OUTCOMES:
Level of epidural catheter insertion: questionnaire | 5 min
  The anesthesiologist will record the intervertebral level at which the epidural was placed: L2-L3, L3-L4
Epidural regimen: questionnaire | 5 min
  Settings for the epidural pump as charted by the anesthesiologist and the nurse.
Maximum upper sensory block to ice: questionnaire | 5 min
  Maximum upper sensory block to ice as charted by the nurse in the electronic charting system
Any anesthetic intervention for patchy or asymmetric block | 5 min
  The anesthetic record will be reviewed for any interventions done.
Number of manual epidural top ups | 5 min
  The number of top ups given by nurses or physicians manually will be recorded from the chart.
Number of PCEA (patient controlled epidural analgesia) boluses delivered | 5 min
  Number of PCEA (patient controlled epidural analgesia) boluses delivered will be collected from the chart.
Duration of epidural analgesia | 5 min
  Time of epidural placement to delivery or placement to top up for caesarean delivery.
Quality of analgesia questionnaire - 1st stage | 5 min
  Quality of analgesia during first stage as defined by the patient on a VNRS (verbal numerical rating scale) 0-10 :
  On a scale from 0-10 (where 0 is not at all and 10 is the best ever), how well did your epidural work from the start of your epidural until you were fully dilated?
Quality of analgesia questionnaire - 2nd stage | 5 min
  Quality of analgesia during second stage as defined by the patient on a VNRS (verbal numerical rating scale) 0-10:
  On a scale from 0-10 (where 0 is not at all and 10 is the best ever), how well did your epidural work from you were fully dilated until the delivery of your baby?

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Bosch OFC, Gleicher Y, Arzola C, Siddiqui N, Downey K, Carvalho JCA. Color flow Doppler in spinal ultrasound: a novel technique for assessment of catheter position in labor epidurals. Reg Anesth Pain Med. 2022 Dec;47(12):775-779. doi: 10.1136/rapm-2022-103948. Epub 2022 Sep 7. PMID 36215115